CLINICAL TRIAL: NCT05446259
Title: Development of a Predictive Outcome Model for Patients With Degenerative Cervical Myelopathy Using Objective Functional and Biological Measures.
Brief Title: Degenerative Cervical Myelopathy Repository
Acronym: DCM
Status: Recruiting | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Francis Farhadi, Associate Professor, University of Kentucky
Other Study IDs: 78340
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Cervical Myelopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood specimens will be collected and banked for future IRB approved research studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DCM group: Subjects diagnosed with degenerative cervical myelopathy.
  Interventions: Other: Standard clinical care procedures and outcome measurements.
- Control group: Subjects diagnosed with cervical spinal disease without myelopathic symptoms.
  Interventions: Other: Standard clinical care procedures and outcome measurements.

INTERVENTIONS:
Other: Standard clinical care procedures and outcome measurements. — Standard of care surgical interventions, imaging impressions, laboratory results, and outcome measurements will be collected and analyzed.

SUMMARY:
To create a research repository of patients with known degenerative cervical myelopathy (DCM) and a control cohort of subjects who have non-myelopathic spinal disease. This repository will be used to assess functional and/or biological measures that may allow for improved prediction of symptomatic progression and response to treatment in patients with DCM. In addition, this repository will be used to develop a risk assessment scale to accurately predict functional outcomes following operative management of DCM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of degenerative cervical myelopathy
* Diagnosis of cervical degenerative disease without myelopathy

Exclusion Criteria:

* None outside or diagnostic requirements and age limits.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be those diagnosed with degenerative cervical myelopathy, and those with cervical degenerative disease who do not experience myelopathic symptoms. Participating subjects will be required to sign the approved informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Data comparison between DCM and control groups | 2 years
  This study is to determine biomarkers associated with DCM and analyze objective clinical measures to determine more predictable and potentially effective treatments for patients diagnosed with cervical myelopathy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided